CLINICAL TRIAL: NCT03215732
Title: Cross Sectional Survey on the Burden and Impacts of Chronic Hepatitis B Virus Infection in the Rural Area of Niakhar, Senegal
Brief Title: Cross Sectional Survey on the Burden and Impacts of Chronic Hepatitis B in the Rural Area of Niakhar, Senegal
Acronym: AMBASS
Status: Completed | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Institute of Research for Development, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS 12356 AMBASS
Record Dates: First submitted 2017-07-10; First posted 2017-07-12 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Chronic Hepatitis b
Keywords: prevalence; vaccine coverage; risk factors; morbidity; mortality; quality of life; economic vulnerability; food security; treatment needs; decentralized care; health costs; caregivers training
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: HBV testing with dried blood spots (DBS) technique — Survey participants will be tested at home for chronic HBV infection using the DBS technique (collection of drops of whole blood dried onto filter paper).

SUMMARY:
This study aims at estimating the prevalence of chronic hepatitis B virus (HBV) infection in rural Senegal (area of Niakhar) and at evaluating the associated burden in terms of both health-related and socio-economic consequences.

DETAILED DESCRIPTION:
The prevalence of chronic HBV infection in Senegal is among the highest worldwide (10% to 17%) but available prevalence estimates relie on studies conducted in specific subgroups (such as military, pregnant women or blood donors).

The prevalence of HBV chronic infection remains undocumented in the general population of Senegal, and its health-related and socio-economic consequences need to be estimated.

This research is based on a cross-sectional survey conducted in the general population with collection of biological, socio-behavioral and economic data at two levels (at the participants' home and in healthcare centers) in the area of Niakhar (located at 135 kms at the East of Dakar).

The research includes three phases as follows:

(i) Preliminary phase: information and communication about the research within the community, training of stakeholders and pilot survey

(ii) Collection of data in the general population

(iii) Communication of results on HBV status to participants and collection of additional data among HBV chronic individuals

ELIGIBILITY:
Inclusion Criteria:

(i) Living in a household of the research zone (individuals living within participating households for at least 6 months, even non permanently: seasonal workers or individuals studying outside the Niakhar zone)

(ii) Being aged of at least 6 months

(iii) Giving informed consent to participate in the research

Exclusion Criteria:

(i) Being an adult unable to sign informed consent

(ii) Being a child whose parents or legal guardian is not present in the household at the time of the survey

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include all individuals who live (even non-permanently) in the sampled households of the Niakhar area for at least 6 months, who are aged of at least 6 months, and who sign informed consent to participate in the survey.
Sampling Method: Probability Sample
Enrollment: 3119 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of chronic HBV infection | At baseline
  HBs Ag positivity with a positive anti-HBc antibody and a negative anti-HBs antibody

SECONDARY OUTCOMES:
Prevalence of chronic HBV infection in age classes '0-15 years; 15-35 years, more than 35 years), and in women of childbearing age | At baseline
  HBs Ag positivity
HBV vaccine coverage (in children born after 2004, year of the introduction of the vaccine in the national program) | At baseline
  HBs Ag negativity with a negative anti-HBc antibody and positive anti-HBs antibody
HBV vaccine efficacy (in children born after 2004, year of the introduction of the vaccine in the national program) | At baseline
  Titration of anti-HBs antibody > 10 UI/l among vaccinated participants
Mortality associated with chronic HBV infection in the Niakhar area | 6 months
  Rate of deaths in the area
Morbidity associated with chronic HBV infection in the Niakhar area | 6 months
  Rate of HBV-related hospitalizations/healthcare use in the area
Quality of life and living conditions of HBV-infected individuals and of their households | 6 months
  Comparison of quality of life scores and socio-economic characteristics between HBV-concerned and HBV not-concerned households
HBV treatment needs in the Niakhar area and in the country | At baseline
  Number of HBV-chronic individuals eligible to HBV treatment (according to WHO criteria) in the area, extrapolation to the needs in other areas of Senegal
Number of quality-adjusted life years(QALYs) lost in the absence of HBV treatment | 6 months
  Use of Markov simulation models
Number of QALYs gained with different scenario of access to HBV treatment | 6 months
  Use of Markov simulation models
Total cost | 6 months
  Use of Markov simulation models (with different scenarii of change in access to HBV treatment and amount of the financial contributions of populations, government and international programs)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie BOYER, Dr, Principal Investigator — Aix Marseille Univ, INSERM, IRD, SESSTIM, Sciences Economiques & Sociales de la Santé & Traitement de l'Information Médicale, Marseille, France
Locations (1):
- At home, Niakhar, Fatick, Senegal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Djaogol T, Perieres L, Marcellin F, Diouf A, Carrieri MP, Diallo A, Boyer S; ANRS 12356 AmBASS Study Group. Hepatitis B prevention and treatment needs in women in Senegal (ANRS 12356 AmBASS survey). BMC Public Health. 2023 May 5;23(1):825. doi: 10.1186/s12889-023-15710-y. PMID 37143029
- [Derived] Coste M, De Seze M, Diallo A, Carrieri MP, Marcellin F, Boyer S; ANRS 12356 AmBASS Study Group. Burden and impacts of chronic hepatitis B infection in rural Senegal: study protocol of a cross-sectional survey in the area of Niakhar (AmBASS ANRS 12356). BMJ Open. 2019 Jul 17;9(7):e030211. doi: 10.1136/bmjopen-2019-030211. PMID 31320358